CLINICAL TRIAL: NCT00687375
Title: A Randomized Controlled Trial of Laparoscopic Inguinal Hernia Repair- Transabdominal Preperitoneal (TAPP) Versus Totally Extra Peritoneal (TEP) Approach
Brief Title: Laparoscopic Inguinal Hernia Repair- Transabdominal Preperitoneal (TAPP) Versus Totally Extra Peritoneal (TEP)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: All India Institute of Medical Sciences (Other)
Responsible Party: Dr. Subodh Kumar, All India Institute of Medical Sciences, New Delhi-29, India
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A-24/2006
Record Dates: First submitted 2008-05-28; First posted 2008-05-30 (Estimated); Last update posted 2008-05-30 (Estimated); Status verified 2008-05

CONDITIONS: Laparoscopic Inguinal Hernia Repair
Keywords: Inguinal; Groin hernia; TAPP; TEP; Comparing; Two; Techniques
MeSH Terms: conditions — Hernia, Inguinal | interventions — tetra-4-amidinophenoxypropane; tetraethylpyrazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Other): Laparoscopic Inguinal Hernia Repair- Transabdominal preperitoneal (TAPP) approach
  Interventions: Procedure: Laparoscopic Inguinal Hernia Repair
- 2 (Other): Laparoscopic Inguinal Hernia Repair- Totally extra peritoneal (TEP) Approach
  Interventions: Procedure: Laparoscopic Inguinal Hernia Repair

INTERVENTIONS:
Procedure: Laparoscopic Inguinal Hernia Repair — Laparoscopic Inguinal Hernia Repair using Transabdominal preperitoneal (TAPP) Approach
  Other Names: TAPP
  Arms: 1
Procedure: Laparoscopic Inguinal Hernia Repair — Laparoscopic Inguinal Hernia Repair using totally extra peritoneal (TEP) Approach
  Other Names: TEP
  Arms: 2

SUMMARY:
Laparoscopic inguinal hernia repair (LIHR) has got comparable results in comparison to open hernia repair (OHR). Many studies have shown that LIHR gives similar results in terms of recurrence as compared with OHR but with the added advantage of less chances of post operative, pain, wound infection and early return to activity. LIHR was started using the transabdominal preperitoneal (TAPP) approach. Another technique of LIHR that has evolved is totally extra peritoneal (TEP) repair. There is only one study of 52 patients comparing TAPP with TEP repair and thus there is insufficient information as to which of the 2 techniques is better. Therefore, we have designed the present study to compare the transabdominal preperitoneal (TAPP) technique with totally extra peritoneal (TEP) technique of laparoscopic inguinal hernia repair. The advantages of TEP may include - no breach of peritoneum so less risk of bowel injury and post-operative adhesions. We will be using a modified technique of TEP repair where we will not use tacker to fix the mesh to reduce the cost of the procedure. On the other hand, TAPP is easy to perform and probably better for irreducible hernia. There is no such comparative study reported in the literature. We have been performing both TAPP and TEP procedures for hernia repair regularly in the department.

RESEARCH HYPOTHESIS: TEP repair of inguinal hernia is better than TAPP repair in terms of reduced cost and avoidance of peritoneal incision.

OBJECTIVE: To compare the Transabdominal preperitoneal (TAPP) vs. Totally extra peritoneal (TEP) techniques of laparoscopic inguinal hernia repair.

DETAILED DESCRIPTION:
The following information from the literature was obtained by searching through the MEDLAR and PUBMED using the key words 'TAPP', 'TEP', 'Laparoscopy' and 'Inguinal hernia'.

Application of laparoscopic techniques has revolutionized the field of surgery. General surgeons have accepted laparoscopic surgery unequivocally. Few would dispute the tremendous success and the impact that laparoscopic cholecystectomy had on the management of gallstone.1 Laparoscopic inguinal hernia repair (LIHR) was introduced following the success of laparoscopic cholecystectomy on the premise that there would be less post-operative discomfort and pain, repair of recurrent hernias would be easier and bilateral hernia can be treated concurrently with improved cosmesis. Ger and Associates2 reported first laparoscopic inguinal hernia repair. Schultz et al3 were the first to report the use of prosthetic material during laparoscopic inguinal hernia repair.

LIHR has got comparable results in comparison to tension free open hernia repair (OHR). Many studies have shown that LIHR gives similar results in terms of recurrence as compared with OHR but with the added advantage of less chances of post operative, pain, wound infection and early return to activity4-6.

Laparoscopic inguinal human repair has undergone tremendous change since its introduction in 1990 by Ger et al3. LIHR was started using the transabdominal preperitoneal (TAPP) approach. TAPP repair involves formation of a peritoneal flap and placement of a mesh in the preperitoneal space. The mesh is then held in place using a tacker. Initially, TAPP became the commonly performed laparoscopic procedure and a number of studies demonstrated the efficacy of TAPP and its comparable results with tension free OHR4-7. Arvidasson D et al8 compared 5 years recurrence rates of laparoscopic inguinal hernia repair Vs. Shouldice repair of primary inguinal hernia which is considered the gold standard for open non-mesh repair of hernia. The cumulative recurrence rate after 5 years was 6.6% in the TAPP group and 6.7% in the Shouldice group. Thus, the TAPP operation represents an excellent alternative to primary inguinal repair.

Wara et al9 have demonstrated that laparoscopic repair compared favourably with Lichteinstein repair for primary indirect and direct hernias, unilateral and bilateral hernias, and recurrent hernias but was inferior for primary bilateral hernias.

Another technique of LIHR that has evolved is totally extra peritoneal (TEP) repair. As the name suggests, the peritoneum is not breached in this technique. Another advantage of TEP repair is that it is not essential to fix the mesh thus avoiding the need for a tacker and bringing down the cost.

There have been 4 non randomized comparative studies that have compared the 2 techniques i.e. TAPP vs TEP (4,10,-12). The results of these comparative trials have shown that the 2 techniques are comparable with regard to the complications such as vascular and visceral injury. However, the port site recurrence was shown to be higher in the TAPP compared with TEP technique. The operating time and the cost of the procedure were not compared in any of the trials.

In a comparative trial of 491 consecutive herniorraphies by Kald et al12, TAPP was compared with TEP. Hernia recurrence was shown to be higher in the TAPP group (7/339 vs 0/87) after a mean follow up of 23(9) and 7(4) months respectively. Other complications were similar with both the techniques (table). However, serious intraabdominal complications occurred in the TAPP group - 2 patients with bowel obstruction and one with severe neuralgion. These complications were not seen with a completely preperitoneal TEP approach. Although the TEP method is technically more difficult, the mean operative time in TAPP (339 patients) and TEP (87 patients) groups were similar {80(32) minutes vs 80 (41) minutes; p = 0.9}. The mean hospital stay and the times to full recovery were also similar in the TAPP and TEP groups. The authors concluded that high quality hernia surgery can be performed with both the TAPP and TEP techniques, but the potential danger of transabdominal route suggests that the TEP operation may be the procedure of choice in laparoscopic inguinal hernia repair.

There is only one randomized controlled trial comparing TAPP with TEP repair13. In this RCT, 52 patients were randomized to either TAPP or TEP. The study showed that the 2 techniques were similar with regard to the complications, time to return to activities and hernia recurrence. However, the length of stay was shorter in the TAPP group (3.7 vs 4.4 days; p=0.03).

TEP repair is preferred for laparoscopic hernia repair because it preserves the peritoneal integrity. However, TEP repair has been associated with a steep learning curve. It's a technically demanding procedure because of the unfamiliar anatomy and requires lot of training and laparoscopic experience. The efficacy of TEP repair as compared to tension free OHR has been studied. It has been found that TEP repair has comparable or even better results than OHR7,14 A gradual shift towards TEP has been observed worldwide because of is advantages such as reduced risk of bowel injury, bowel adhesions and incisional hernia formation.

However, since there is only one RCT involving only 52 patients, the Cochrane database review 200511 has concluded that there are insufficient data comparing TAPP and TEP techniques of laparoscopic inguinal hernia repair.

Therefore, we have designed the present study to compare the transabdominal preperitoneal (TAPP) technique with totally extra peritoneal (TEP) technique of laparoscopic inguinal hernia repair. We will be using a modified technique of TEP repair where we will not use tacker to fix the mesh reduce the cost of the procedure. There is no such comparative study reported in the literature.

We have been performing both TAPP and TEP procedures for hernia repair in the department. Both these procedures are well standardized.

PATIENTS AND METHODS

Study Design: Prospective randomized controlled trial. Selection of cases and inclusion criteria: All consecutive patients with uncomplicated symptomatic inguinal hernia attending the out patient department of surgery at AIIMS will be included in the study. The diagnosis of inguinal hernia will be made clinically.

Exclusion criteria: Patients will be excluded if there is - (i) Co-morbid conditions making the patients unfit for general anesthesia (ii) Complicated hernia. (iii) Uncorrectable coagulopathy (iv) Morbid obesity (Body Mass Index > 30) (v) Suspected intra-abdominal or pelvic malignancy.

METHODS: All patients with uncomplicated inguinal hernia planned for laparoscopic inguinal hernia repair will be randomized to receive either TAPP or TEP technique for hernia repair. Randomization will be done by using random number table.

Pre-operative Preparation: Single dose of injection Amoxycillin 1000mg + Clavulinic acid 250mg AST i.v. will be given as prophylaxis preoperatively. Part will be shaved and cleaned properly. Patient will be catheterized before the start of the procedure.

Operative Procedure

General Anesthesia- Patient will be placed in supine position with both upper limbs by the side of the patient. Induction will be done by propofol and maintenance by O2+N2O+Isoflurane and vecuronium. Patients will be kept on intermittent positive pressure ventilation during the procedure.

Technique of TAPP repair:

Pneumoperitoneum upto 14 mmHg will be created with CO2 using Veress needle at umbilicus. A standard 10 mm trocar will be placed 1 cm below the umbilicus for insertion of laparoscope. Two additional 5 mm trocars will be placed at the same level approximately 5-6 cm on either side of the umbilicus. The contents of the inguinal hernia (if any) will be pulled back into the abdomen. A short curved incision will be made lateral to the inguinal ring extending transversely below the semilunar line, to enable the formation of a peritoneal flap until the identification of the inferior epigastric vessels medially. The rectus muscle will be used to identify the pubic tubercle and Cooper's ligament.

After the dissection, a rolled piece of polypropylene mesh (10x15 cm) will be introduced via umbilical port into the abdomen. After unrolling the mesh, it will cover the entire inguinal area on the affected side. No tacker will be used to fix the mesh. The peritoneal flaps will be closed back to cover the mesh completely using absorbable suture 2-0 polydiaoxanon (PDS); this is to prevent adhesions between mesh and intestine. The CO2 will be released, the midline trocar fascia will be closed, and then the other trocar sites will be closed with simple suture using 3-0 nylon.

Technique of TEP Procedure:

All three ports will be made in the midline. A 10 mm port just below the umbilicus will be made for telescope. The rectus muscle will be retracted laterally after incising the rectus sheath and a blunt dissection done using the balloon dissector or telescope to create preperitoneal space until the pubis is felt. Two 5 mm ports will be made, one just above the pubis and the other in the midline between 10 mm port and 5 mm pubis port. The entire posterior floor will be dissected and the anatomical landmarks recognized. A single sheet of mesh will be introduced. It the peritoneum or hernial sac gets inadvertently opened during dissection, it will be sutured or ligated with a chromic endoloop, if possible. The mesh will be left in the preperitoneal space adequately covering the deep inguinal ring, Hasselback's triangle and femoral hernia site. No tacker will be used to fix the mesh. The CO2 will be released. The 10 mm port fascia will be closed using 1-0 vicryl, and then the 5mm port sites will be closed with simple suture using 3-0 nylon.

Any intra-operative complications like vascular, nerve or vas injury, peritoneal breach and serious visceral injuries will be recorded. The operative time will be recorded as the time from the incision until the last skin stitch. Any conversions from totally extra peritoneal technique to transabdominal preperitoneal technique and from laparoscopic to open repair will be recorded with the specific reason for conversion. The ease of operation will be graded as - easy / moderately difficult / difficult.

Bleeding will be recorded as mild if no suction irrigation is required, moderate if suction is required at the end of the procedure or if suction is required to improve vision, and severe if blood transfusion is required.

For postoperative pain relief, injection diclofenac sodium 75 mg i.m. and for vomiting injection ondansetron 8 mg i.v. will be given post-operatively in the recovery room to all patients. Pain will be recorded at 1, 6, 24 hours after operation, at the time of discharge and during follow up on a Visual Analogue Scale (VAS) with end points labeled as no pain and worst possible pain on a scale of 10.

Visual analogue scale No pain Worst possible pain

0 1 2 3 4 5 6 7 8 9 10

_____________________________________________________________

Extra analgesic and antiemetic requirements, post-operative time to resume feeding, return of bowel activity, total hospital stay, any urinary retention will be the other variables measured post-operatively.

Complications including haematoma / seroma formation and wound infections will be recorded. The port site wound infections will be classified according to the CDC classification for surgical site infection15 :

1. Superficial incisional - involving only skin and superficial tissue i.e. subcutaneous tissue.
2. Deep incisional - involving fascial and muscle layer.
3. Organ/space infection - involving any part of anatomy, other than incision which is opened or manipulated e.g. post-operative intraabdominal abscess.

Recurrence and cosmesis will be recorded during follow-up. Cosmesis will be analyzed by patient's satisfaction score on surgery and on scar, which will be labeled on verbal rating scale (VRS) with score of:

0 = Not satisfied

1. = Partially satisfied
2. = Satisfied
3. = Very satisfied

ELIGIBILITY:
Inclusion Criteria:

* All consecutive patients with uncomplicated symptomatic inguinal hernia attending the out patient department of surgery at AIIMS will be included in the study.
* The diagnosis of inguinal hernia will be made clinically.

Exclusion Criteria:

* Co-morbid conditions making the patients unfit for general anaesthesia
* Complicated hernia.
* Uncorrectable coagulopathy
* Morbid obesity (Body Mass Index > 30)
* Suspected intra-abdominal or pelvic malignancy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2007-04; Primary Completion 2008-05 (Estimated); Study Completion 2009-03 (Estimated)

PRIMARY OUTCOMES:
Operating time (in minutes) | Two years
Cost of the procedure | Two years

SECONDARY OUTCOMES:
Conversion rate | Two years
Recurrence of hernia | Two years
Major complications | Two years

CONTACTS AND LOCATIONS:
Overall Officials: Subodh Kumar, MBBS, MS, Principal Investigator — All India Institute of Medical Sciences, New Delhi-29, India
Locations (1):
- All India Institute of Medical Sciences, New Delhi, New Delhi, National Capital Territory of Delhi, India